CLINICAL TRIAL: NCT06061991
Title: Mobile Instant Messaging-based Lifestyle Interventions for Preventing Gestational Diabetes in High-risk Pregnant Women: a Randomised Controlled Trial
Brief Title: Mobile Instant Messaging-based Lifestyle Intervention for Gestational Diabetes Prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Tzu Tsun Luk, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17101423
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gestational Diabetes
Keywords: lifestyle modification; gestational weight gain; Chinese; digital health; mHealth; WhatsApp
MeSH Terms: conditions — Diabetes, Gestational; Gestational Weight Gain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Mobile instant messaging-based lifestyle intervention
  Interventions: Behavioral: Mobile instant messaging-based lifestyle intervention; Behavioral: Brief advice on GDM prevention; Behavioral: Usual care
- Control group (Active Comparator): Brief advice on GDM prevention
  Interventions: Behavioral: Text messaging reminders; Behavioral: Brief advice on GDM prevention; Behavioral: Usual care

INTERVENTIONS:
Behavioral: Mobile instant messaging-based lifestyle intervention — Nurse-led personalised lifestyle intervention grounded in social cognitive theory via WhatsApp or WeChat from baseline to the 28th gestational week, which aims to maintain optimal gestational weight gain using dietary and exercise advice and behavioural change techniques.
  Arms: Intervention group
Behavioral: Text messaging reminders — Follow-up reminders via text messaging as attention control.
  Arms: Control group
Behavioral: Brief advice on GDM prevention — Brief advice on GDM prevention aided by an A4-sized, half-fold leaflet, which covered the risk factors and complications of GDM, optimal gestational weight gain targets, and advice on dietary and exercise during pregnancy
Behavioral: Usual care — Usual care provided by the prenatal clinic.

SUMMARY:
The goal of this randomised controlled trial is to test the effectiveness of a mobile instant messaging-based lifestyle intervention in pregnant women at risk of gestational diabetes

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is one of the most common medical conditions during pregnancy, affecting about 1 in 7 live births worldwide. There remains a lack of proven preventive strategies for GDM that could be readily adopted in clinical practice. Recent studies have suggested that lifestyle intervention delivered via mobile phone could help pregnant women prevent GDM, but more evidence is needed. This study aims to test a mobile instant messaging-based lifestyle intervention for GDM prevention in pregnant women at risk of GDM.

ELIGIBILITY:
Inclusion Criteria:

1. Ethnic Chinese singleton pregnant woman in <14 weeks of gestation
2. Aged 18 years or above
3. Own a mobile phone with an instant messaging app
4. Not participating in similar trials on diabetes or lifestyle modifications
5. Have at least one of the following risk factors for GDM:

   * Age ≥35 years at the expected date of delivery
   * Body mass index (BMI) ≥ 25 kg/m2 pre-pregnancy or in the first trimester
   * Family history of diabetes in first-degree relative
   * Previous GDM or delivered a baby with birthweight ≥4 kg

Exclusion Criteria:

* Pre-existing diabetes or other medical conditions that may affect metabolism (e.g., thyroid disorders) or psychiatric disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 944 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
GDM diagnosis | About 28th gestational week
  GDM diagnosed by a 2-hour 75g oral glucose tolerance test interpreted according to the World Health Organization's 2013 criteria

SECONDARY OUTCOMES:
Gestational weight gain | From baseline to the end of pregnancy (delivery)
  Measured in kilograms
Hypertensive disorders of pregnancy | During pregnancy
  Including gestational hypertension and preeclampsia
Pharmacological therapy for hyperglycaemia | During pregnancy
  Such as metformin and insulin
Mode of birth | At delivery
  Such as normal spontaneous delivery, caesarean section, assisted vaginal delivery
Gestational age at birth | At delivery
  Measured in weeks and days
Birthweight | At birth
  Measured in grams
Large for gestational age | At birth
Small for gestational age | At birth
Preterm birth | At birth
  Defined as birth before the 37th gestational week
Neonatal hypoglycaemia | At birth
Neonatal death | Within 28 days after birth
  Defined as death within 28 days after birth
Stillbirth | During pregnancy
  Defined as fetal death after the 20th gestational week

CONTACTS AND LOCATIONS:
Overall Officials: Tzu Tsun Luk, PhD, RN, Principal Investigator — The University of Hong Kong
Locations (4):
- Hong Kong (4):
  - Kwong Wah Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital/ Tsan Yuk Hospital, Hong Kong
  - United Christian Hospital/ Tseung Kwan O Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No